CLINICAL TRIAL: NCT00693381
Title: An Open, Multicentre, Randomised, Parallel Group Pilot-Study to Compare Safety and Efficacy of Discontinuation of Mycophenolate Mofetil From a Tacrolimus/MMF/Steroid Triple Regimen Following Kidney Transplantation
Brief Title: Mycophenolate Mofetil (MMF) Discontinuation From a Tacrolimus/MMF/Steroid Triple Regimen After Kidney Transplantation
Acronym: DISTAMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-02-CEE-01
Record Dates: First submitted 2008-06-03; First posted 2008-06-09 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Kidney Transplantation
Keywords: Transplantation; Graft Rejection; Renal Transplantation
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Methylprednisolone; Prednisone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tacrolimus/MMF/steroids throughout the study
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: methylprednisolone and prednisone
- 2 (Experimental): Tacrolimus/MMF/steroids with MMF reduction from week 7 to 12 and MMF discontinuation at month 3
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: methylprednisolone and prednisone

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: Prograf; FK506
Drug: Mycophenolate Mofetil — oral
  Other Names: CellCept
Drug: methylprednisolone and prednisone — IV and oral
  Other Names: Steroids

SUMMARY:
Patients after kidney transplantation received immunosuppression by Tacrolimus, MMF and steroids. In one half of the patients after 7 weeks MMF was reduced by half, and after 12 weeks it was stopped. For the others MMF remained at initial dose.

ELIGIBILITY:
Inclusion Criteria:

* Patient has an end stage kidney disease and is a suitable candidate for primary renal transplantation or retransplantation
* Patient is receiving a kidney transplant, from a cadaveric or living donor between 5 and 65 years of age with compatible ABO blood type

Exclusion Criteria:

* Patient has an immunological high risk, defined as having a most recently measured PRA grade of >= 50% within the previous six months
* Patient requires ongoing dosing with a systemic immunosuppressive drug at study entry for any reason other than kidney transplantation
* Patient requires initial sequential or parallel therapy with immunosuppressive antibody preparation(s)
* Patient or donor is known to be HIV positive
* Patient with malignancy or history of malignancy, except non metastatic basal or squamous cell carcinoma of the skin that has been treated successfully
* Patient has significant, uncontrolled concomitant infections and/or severe diarrhoea, vomiting, or active peptic ulcer
* Patient is receiving a graft from a non-heart-beating donor
* Cold ischemia time of the donor kidney >= 40 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2003-02; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Incidence of and time to first biopsy proven acute rejection over the first 6 months post transplantation | 6 months

SECONDARY OUTCOMES:
Incidence and seriousness of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (14):
- Czechia (4):
  - Brno
  - Hradec Králové
  - Olomouc
  - Ostrava
- Hungary (2):
  - Debrecen
  - Pécs
- Poland (7):
  - Bialystok
  - Gdansk
  - Krakow
  - Lublin
  - Warsaw
  - Wroclaw
  - Zabrze
- Banska, Slovakia

REFERENCES:
- [Background] Sulowicz W, Bachleda P, Rydzewski A, Rutkowski B, Szakaly P, Asztalos L, Samlik J, Lackova E, Ksiazek A, Studenik P, Mysliwiec M, Hruby Z, Navratil P, Gumprecht J. Discontinuation of mycophenolate mofetil from a tacrolimus-based triple regimen 2 months after renal transplantation: a comparative randomized, multicentre study. Transpl Int. 2007 Mar;20(3):230-7. doi: 10.1111/j.1432-2277.2006.00421.x. PMID 17291216